CLINICAL TRIAL: NCT05873959
Title: An Observational Multicenter Study to Evaluate the Safety and Efficacy of Humacyte's Human Acellular Vessel in a Real World Setting for Arterial Replacement or Reconstruction in Ukrainian Patients With Life or Limb-threatening Vascular Trauma
Brief Title: An Observational Study to Evaluate the Safety and Efficacy of Humacyte's HAV for Arterial Replacement or Reconstruction in Ukrainian Patients With Life or Limb-threatening Vascular Trauma
Status: Completed | Type: Observational
Sponsor: Humacyte, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-PRO-V017
Expanded Access: NCT03631056 (Approved for marketing)
Record Dates: First submitted 2023-05-16; First posted 2023-05-24 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Trauma; Trauma Injury; Trauma, Multiple; Trauma Blunt
Keywords: extremities; arterial replacement; arterial reconstruction
MeSH Terms: conditions — Wounds and Injuries; Accidental Injuries; Multiple Trauma; Wounds, Nonpenetrating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: HAV implantation — HAVs already implanted under humanitarian aid program to repair or reconstruct arteries following an extremity life- or limb-threatening traumatic injury.

SUMMARY:
Humacyte provided HAVs as humanitarian aid to Ukraine. This retrospective observational study is designed to collect data from patients in whom the HAVs have already been implanted on a humanitarian basis between June 2022 and May 2023.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an HAV implanted to repair or reconstruct an arterial vessel following life- or limb-threatening traumatic vascular injury of an extremity.
* Aged 18 to 85 years old, inclusive.
* Patient or legal representative is able, willing, and competent to give informed consent.

Exclusion Criteria:

• Employees of the sponsor or patients who are employees or relatives of the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with vascular trauma in the extremities who required arterial replacement or reconstruction and in whom the HAVs have been already implanted on a humanitarian basis between June 2022 and May 2023.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of the HAV | up to 12 months
  To determine the rate of adverse events after impanation
Primary patency of the HAV after implantation | 30 days
  To determine the rate of HAV primary patency at 30 days after implantation

SECONDARY OUTCOMES:
Frequency of Adverse Events of Special Interest (AESIs) | up to 12 months
  To determine the rate of Adverse Events of Special Interest (AESIs), such as: thrombosis, clinically significant aneurysm or pseudoaneurysm formation, HAV spontaneous rupture, infection of the HAV conduit, and HAV abandonment.
HAV durability | up to 12 months
  To determine the time frame when the HAV has not been removed, replaced, or ligated.
Rate of affected limb salvage/amputation after implantation | up to 12 months
  To determine the rate of affected limb salvage/amputation after HAV implantation
Patency of the HAV after implantation | up to 12 months
  To determine the rate of HAV patency (primary, primary assisted, and secondary) after implantation

CONTACTS AND LOCATIONS:
Locations (3):
- Ukraine (3):
  - Municipal Non-Profit Enterprise ""City Clinical Hospital #16" of the Dnipro City Council", Dnipro
  - Medical Center LLC "CLINIC VERUM EXPERT", Kyiv
  - Communal non-profit enterprise "Vinnytsia Regional Clinical Hospital named after E. Pirogov" of the Vinnytsia Regional Council, center of cardiovascular surgery, Vinnytsia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sokolov O, Shaprynskyi V, Skupyy O, Stanko O, Yurets S, Yurkova Y, Niklason LE. Use of bioengineered human acellular vessels to treat traumatic injuries in the Ukraine-Russia conflict. Lancet Reg Health Eur. 2023 May 6;29:100650. doi: 10.1016/j.lanepe.2023.100650. eCollection 2023 Jun. No abstract available. PMID 37213923
- [Result] Moore EE, Curi M, Namias N, Kundi R, Lum YW, Fox CJ, Rajani RR, Rasmussen TE, Sokolov O, Niklason LE, Khondker Z, Parikh SJ; CLN-PRO-V005 Investigators and the CLN-PRO-V017 Investigators. Bioengineered Human Arteries for the Repair of Vascular Injuries. JAMA Surg. 2025 Feb 1;160(2):181-189. doi: 10.1001/jamasurg.2024.4893. PMID 39565635
- See also: Lancet Regional Health Europe — https://doi.org/10.1016/j.lanepe.2023.100650